CLINICAL TRIAL: NCT00716781
Title: Management of Infants Born to Group B Streptococcus Positive Mothers: Laboratory Tests vs Physical Examination
Brief Title: Management of Infants Born to Group B Streptococcus Positive Mothers.
Status: Completed | Type: Observational
Sponsor: IRCCS Burlo Garofolo (Other)
Collaborators: Friuli Venezia Giulia Regional Health Authority (Unknown)
Responsible Party: Sergio De Marini, IRCCS Burlo Garofolo
Other Study IDs: GBS FVG 2004-2006
Record Dates: First submitted 2008-07-14; First posted 2008-07-16 (Estimated); Last update posted 2008-07-16 (Estimated); Status verified 2008-07

CONDITIONS: Group B Streptococcus; Sepsis; Infant, Newborn
Keywords: Group B streptococcus; Sepsis; Infants; Diagnosis; Physical examination; Laboratory tests
MeSH Terms: conditions — Sepsis; Disease

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1 (first year): Asymptomatic infants born to GBS-positive mothers or to mothers with risk factors and incomplete prophylaxis were managed according to the CDC protocol. Blood cultures and CBC were performed and the infant was observed for 48 hours. Participating hospital were free to perform any additional test, such as CRP, MiniESR, etc
- 2 (second year): Asymptomatic infants born to GBS-positive mothers or to mothers with risk factors and incomplete prophylaxis were managed with clinical observation only. Clinical surveillance was based on 3 signs: 1. Skin appearance (pink, pale, mottled, cyanotic); 2. Respiratory rate (>50 or <50 breaths per minute); 3. Dyspnea (Yes / No)

SUMMARY:
Intrapartum antibiotic prophylaxis has greatly decreased but not abolished early-onset neonatal sepsis caused by GBS. According to current recommendations, the evaluation of infants at risk for GBS sepsis should include a complete blood count (CBC), WBC differential, a blood culture (BC) and a period of observation. The usefulness of CBC and BC in the evaluation process is not firmly established.

DETAILED DESCRIPTION:
After implementation of appropriate guidelines, early-onset GBS sepsis has become a low incidence disease (CDC). Recent rates are as low as 0.34 cases /1000 live births. According to CDC recommendations, the evaluation of infants at risk for GBS sepsis should include a complete blood count (CBC), WBC differential, a blood culture (BC) and a period of observation. The usefulness of CBC and BC in the evaluation process is not firmly established. There are several reviews on the predictive value of CBC and putative markers of early onset neonatal sepsis, but there seems to be no ideal laboratory test to assist the clinician in the diagnosis (Fowlie 1998, Malik 2003, Ottolini 2003). Given the continuing concerns about the reliability of laboratory tests, one may ask the question of whether physical examination might be at least as good as haematological indices. We are not aware of studies assessing the value of physical examination vs CBC, in the evaluation of asymptomatic at risk newborns.

The aim of this study was to compare two approaches in the management of infants at risk for GBS sepsis: laboratory tests (CBC, differential and BC) with observation vs clinical observation alone.

ELIGIBILITY:
Inclusion Criteria:

* All newborns born in Friuli Venezia Giulia Region (Italy)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All newborns born in Friuli Venezia Giulia Region (Italy) during the study period
Sampling Method: Non-Probability Sample
Enrollment: 16394 (Actual)
Dates: Start 2004-07; Primary Completion 2006-06 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Number of infants treated with antibiotics | Study period

SECONDARY OUTCOMES:
Time elapsed from the onset of symptoms to the beginning of antibiotic treatment | Study period

CONTACTS AND LOCATIONS:
Overall Officials: Sergio De Marini, MD, Study Chair — IRCCS Burlo Garofolo, Trieste, Italy; Luigi Cantoni, MD, Principal Investigator — San Daniele Hospital, San Daniele, Italy

REFERENCES:
- [Derived] Cantoni L, Ronfani L, Da Riol R, Demarini S; Perinatal Study Group of the Region Friuli-Venezia Giulia. Physical examination instead of laboratory tests for most infants born to mothers colonized with group B Streptococcus: support for the Centers for Disease Control and Prevention's 2010 recommendations. J Pediatr. 2013 Aug;163(2):568-73. doi: 10.1016/j.jpeds.2013.01.034. Epub 2013 Mar 8. PMID 23477995